CLINICAL TRIAL: NCT03960203
Title: Effect of a Sepsis Prediction Algorithm on Patient Mortality, Length of Stay, and Readmission
Brief Title: Effect of a Sepsis Prediction Algorithm on Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dascena (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Diagnostic
Other Study IDs: 05172019
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Severe Sepsis
Keywords: Dascena; Patient mortality; Length of stay; Readmissions; Algorithm; Diagnostic; Clinical outcomes
MeSH Terms: conditions — Sepsis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparator (Experimental): The comparator arm will involve patients monitored by InSight.
  Interventions: Diagnostic Test: InSight

INTERVENTIONS:
Diagnostic Test: InSight — Clinical decision support (CDS) system for severe sepsis detection and prediction

SUMMARY:
In this clinical outcomes analysis, the effect of a machine learning algorithm for severe sepsis prediction on in-hospital mortality, hospital length of stay, and 30-day readmission was evaluated.

DETAILED DESCRIPTION:
Materials and Methods: Clinical outcomes evaluation performed on a multiyear, multicenter clinical data set of real-world data containing 75,147 patient encounters from nine hospitals. Mortality, hospital length of stay, and 30-day readmission analysis performed for 17,758 adult patients who met two or more Systemic Inflammatory Response Syndrome (SIRS) criteria at any point during their stay.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 presenting to the emergency department or admitted to an inpatient unit at the participating facilities were automatically included for clinical outcomes analysis

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75147 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 1 year
  Rate of in-hospital mortality based on SIRS criteria

SECONDARY OUTCOMES:
Hospital length of stay | 1 year
  Duration of hospital length of stay in days based on SIRS criteria
30-day readmissions | 1 year
  Rate of patient readmissions within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ritankar Das, MSc, Principal Investigator — Dascena

REFERENCES:
- [Derived] Burdick H, Pino E, Gabel-Comeau D, McCoy A, Gu C, Roberts J, Le S, Slote J, Pellegrini E, Green-Saxena A, Hoffman J, Das R. Effect of a sepsis prediction algorithm on patient mortality, length of stay and readmission: a prospective multicentre clinical outcomes evaluation of real-world patient data from US hospitals. BMJ Health Care Inform. 2020 Apr;27(1):e100109. doi: 10.1136/bmjhci-2019-100109. PMID 32354696